CLINICAL TRIAL: NCT05040555
Title: A Prospective Clinical Study of R-CDOP Regimen in the Treatment of Newly Diagnosed Non-Hodgkin's Lymphoma With High Tumor Burden
Brief Title: R-CDOP Regimen in the Treatment of Newly Diagnosed Non-Hodgkin's Lymphoma With High Tumor Burden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: oubai, MD/PhD (Other)
Responsible Party: Sponsor-Investigator, oubai, MD/PhD, Director, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-NHL-001
Record Dates: First submitted 2021-08-31; First posted 2021-09-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma Grade 3B
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CDOP (Experimental): Rituximab 375mg/m2, D0; Cyclophosphamide 750mg/ m2, D1; Doxorubicin hydrochloride liposome 30-35mg/ m2, D1; Vindesine 3mg/ m2, D1; Prednisone 60mg/ m2, D1~5.
  Interventions: Combination Product: R-CDOP

INTERVENTIONS:
Combination Product: R-CDOP — Rituximab 375mg/m2, D0; Cyclophosphamide 750mg/ m2, D1; Doxorubicin hydrochloride liposome 30-35mg/ m2, D1; Vindesine 3mg/ m2, D1; Prednisone 60mg/ m2, D1~5.

SUMMARY:
A single-center, prospective clinical study to evaluate the efficacy and safety of R-CDOP (Rituximab, Cyclophosphamide, Doxorubicin hydrochloride liposome, Vindesine, Prednisone ) in the treatment of newly diagnosed high tumor burden non-Hodgkin's lymphoma, which has previously shown promising efficacy.

DETAILED DESCRIPTION:
The objective was to evaluate the efficacy and safety of R-CDOP regimen in the initial treatment of Patients with at least one of the following high tumor burden, and to provide a basis for the application of Doxorubicin hydrochloride liposome.

At least 3 nodal sites (each with a diameter greater than 3 cm) ; Nodal or extranodal mass > 7cm in its greater diameter; Hepatomegaly and splenomegaly (infiltration confirmed by PET-CT; Spleen: female > 15cm, male > 16cm) ; Pleural/peritoneal effusion; Lactate dehydrogenase (LDH) three times the upper limit of normal; PET-CT Total Metabolic Tumor Volume (TMTV)>220cm3.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically immunohistochemistry and imaging confirmed diffuse large B-cell lymphoma or follicular lymphoma grade 3B;
2. Has at least one evaluable or measurable lesion according to Lugano response criteria;
3. Patients with at least one of the following high tumor burden Involvement of at least 3 nodal sites (each with a diameter greater than 3 cm); nodal or extranodal mass > 7cm in its greater diameter; Hepatomegaly and splenomegaly (infiltration confirmed by PET-CT; Spleen: female > 15cm, male > 16cm); Pleural/peritoneal effusion; Lactate dehydrogenase (LDH) three times the upper limit of normal; PET-CT TMTV >220cm3;
4. Patients previously untreated;
5. Patients aged over 18 and under 75 years;
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0~2;
7. International Prognostic Index (IPI) score > 1, or with extranodal mass diameter ≥7cm;
8. Life expectancy ≥ 6 months;
9. Left Ventricular Ejection Fraction (LVEF) ≥ 50%;
10. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Pregnant or lactation and patients of childbearing age who do not want to take contraceptive measures;
2. Abnormal liver function [total bilirubin > 1.5 times of the upper limit of normal value; Alanine aminotransferase/Aspartate aminotransferase (ALT / AST) > 2.5 times of upper limit of normal value for patients without liver metastasis ; ALT / AST > 5 times of upper limit of normal value for patients with liver metastasis ], abnormal renal function (serum creatinine > 1.5 times of upper limit of normal value) ;
3. Absolute Neutrophil Count (ANC)<1.5×10^9/L or Platelet (PLT)< 75 × 10^9/L;
4. Hypersensitivity to any study drug or its ingredients;
5. Patients with significant and uncontrolled cardiovascular disease or history;
6. Persons with mental disorders/unable to obtain informed consent;
7. Lymphoma infiltrates the central nervous system;
8. Previous history of malignant tumor;
9. HIV infection; HBV infection (HBV-DNA> 2000 IU/ml);HCV infection (HCV-RNA>200 IU/ml);
10. The investigator determined not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Percentage of Complete remission (CR), and Partial remission (PR), referred to Lugano 2014.

SECONDARY OUTCOMES:
Disease Control Rate | 24 months
  Percentage of Complete remission (CR), Partial remission (PR), and stable disease (SD), referred to Lugano 2014.
Progression-free survival | 24 months
  Progression-free survival（PFS） is defined as the time from the date of enrollment to the date of first documentation of progressive disease (PD) or death from any cause.
Overall survival | 60 months
  Overall survival（OS） is defined as the time from the date of enrollment to the date of death from any cause.
Adverse Events | 24 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No